CLINICAL TRIAL: NCT03737578
Title: Efficacy of Daily Hemodialysis Compared With in Center Hemodialysis 3 Times Per Week
Brief Title: Comparison of Daily Home Hemodialysis (HD) With Conventional in Center HD in Terms of Patients Quality of Life and Clinical Outcomes
Acronym: SeCoIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Physidia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018A00838-47
Record Dates: First submitted 2018-10-22; First posted 2018-11-09 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: End Stage Renal Disease
Keywords: Home hemodialysis; Daily hemodialysis; Frequent hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: this is an interventional, pragmatic study with minimal risks, exposed / unexposed, prospective, longitudinal, multicentric and national conducted in metropolitan France
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily hemodialysis patients (Experimental): Description: End stage renal disease patients starting daily hemodialysis treatment.
  Interventions: Delivery of a connected pedometer / accelerometer and Quality Of Life and Restless Leg Syndrome questionnaires.
  Interventions: Other: Delivery of a connected pedometer / accelerometer
- Conventional hemodialysis patients (Active Comparator): Description: End stage renal disease patients currently treated by conventional hemodialysis or starting conventional hemodialysis treatment.
  Interventions: Delivery of a connected pedometer / accelerometer and Quality Of Life and Restless Leg Syndrome questionnaires.
  Interventions: Other: Delivery of a connected pedometer / accelerometer

INTERVENTIONS:
Other: Delivery of a connected pedometer / accelerometer — Delivery of a connected pedometer / accelerometer that the patient will be asked to wear at least 7 consecutive days / month.
  Quality of life and leg restless syndrome questionnaires (auto questionnaire) completed by the patients every 3 months
  Other Names: Quality of life and restless leg syndrome questionnaires

SUMMARY:
The objective of this study is to describe the characteristics of patients on daily home hemodialysis and to confirm in real practice in France the effectiveness shown in studies, mainly American, both in terms of clinical outcomes and quality of life. Due to the few studies available in this population, the focus will be particularly on physical activity.

DETAILED DESCRIPTION:
Primary objective :

The main objective of this study is to evaluate the physical activity in the daily life of patients in daily hemodialysis in comparison with patients treated 3 times a week (conventional hemodialysis) others objectives are also:

1. To describe the characteristics of daily hemodialysis patients;
2. To describe the prescription procedures of the home daily HD;
3. To compare the evolution of the blood pressure between the 2 modalities of hemodialysis;
4. To compare the frequency of hospitalizations, duration and hospitalization reasons between the 2 hemodialysis modalities;
5. To compare the quality of life of the patients between the 2 modalities ;
6. To evaluate the quality of the sleep of the patients between the 2 modalities ;
7. Compare the percentage of patients with restless leg syndrome (RLS) and the severity of RLS between the two modalities;
8. Compare the evolution of drug intake between the two modalities;
9. Evaluate the number of abandoning subjects and causes of discontinuation of HQD;

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or over
2. Patient who dated and signed the consent form
3. Patient (s) affiliated to a Social Security scheme
4. Interventional arm: patient who begins or will begin daily hemodialysis training (5, 6 or 7 times per week) at home.
5. Comparator arm: prevalent or incident patient treated by conventional hemodialysis (3 times per week) and fitting with the matching criteria of an interventional patient included in the center

Exclusion Criteria:

1. Patient with needs any help to walk (wheelchair, crutch, walker, cane ...)
2. Patient with active neoplasia;
3. Patient with predicted life expectancy of less than one year;
4. Patient with significant reading or writing difficulties;
5. Patient participating in a clinical trial or other interventional study; 6. Patient with history of mental instability, major cognitive impairment in the previous 5 years, or major psychiatric condition not adequately controlled or stable under pharmacological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Physical activity of patients (total average number of steps taken per day through connected pedometer/accelerometer) | 3 months
  The main criteria is the total average number of steps taken per day
Physical activity of patients (total average number of steps taken per day through connected pedometer/accelerometer) | 6 months
  The main criteria is the total average number of steps taken per day
Physical activity of patients (total average number of steps taken per day through connected pedometer/accelerometer) | 9 months
  The main criteria is the total average number of steps taken per day
Physical activity of patients (total average number of steps taken per day through connected pedometer/accelerometer) | 12 months
  The main criteria is the total average number of steps taken per day

SECONDARY OUTCOMES:
Evolution of the blood pressure during the study period | At inclusion and during visit at month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Systolic and diastolic blood pressure measurement
Evolution of the frequency of hospitalizations during the study period | During visit at month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  number of hospitalizations period
Change in quality of life of the patients measured through questionnaire during the study period | At inclusion and during visit at month 3, 6, 9 and 12
  Questionnaire KDQOL-SF version 1.2 (auto questionnaire)
Change in quality of the sleep of the patients through questionnaire during the study period | At inclusion and during visit at month 3, 6, 9 and 12
  Pittsburgh Sleep Quality Index PSQI version 1.0 (auto questionnaire)
Change of the percentage of patients with restless leg syndrome (RLS) during the study period | At inclusion and during visit at month 3, 6, 9 and 12
  International scale of Restless leg syndrome severity IRLS V1.0 (auto questionnaire)
Change of drug intake during the study period (posology of drugs linked with ESRD) | During visit at month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Evolution of drugs posology (drug linked with ESRD)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Target, MD, Principal Investigator — Centre Hospitalier La Roche sur Yon - France; Cécile Courivaud, MD, Study Chair — CHRU Jean Minjoz, Besançon, France; Pierre Antoine Michel, MD, Study Chair — Hôpital Tenon APHP, Paris, France
Locations (1):
- Centre Hospitalier, La Roche-sur-Yon, France

REFERENCES:
- [Derived] Target N, Courivaud C, Michel PA, Daoud S, Thomas M. Comparison of physical activity and quality of life in home haemodialysis (HHD) patients versus conventional in-centre haemodialysis (ICHD) patients: the observational, longitudinal, prospective, international, multicentric SeCoIA study protocol. BMC Nephrol. 2020 Nov 23;21(1):500. doi: 10.1186/s12882-020-02127-7. PMID 33225917